CLINICAL TRIAL: NCT05423951
Title: Effect of Remimazolam and Propofol on Hemodynamic Stability During Anesthesia Induction in Patients Undergoing Coronary Artery Bypass Grafting
Brief Title: Effect of Remimazolam and Propofol on Hemodynamic Stability During Anesthesia Induction in OPCAB Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Remimazolam_OPCAB
Record Dates: First submitted 2022-06-12; First posted 2022-06-21 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Hemodynamic Instability
Keywords: hemodynamics; remimazolam; propofol; coronary artery bypass grafting
MeSH Terms: interventions — Injections, Intravenous; Powders; Propofol; Rocuronium; Sufentanil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental)
  Interventions: Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO]; Drug: Rocuronium; Drug: Sufentanil
- Propofol (Active Comparator)
  Interventions: Drug: Propofol; Drug: Rocuronium; Drug: Sufentanil

INTERVENTIONS:
Drug: REMIMAZOLAM BESYLATE 2.5 Mg in 1 mL INTRAVENOUS INJECTION, POWDER, LYOPHILIZED, for SOLUTION [BYFAVO] — For the induction of anesthesia, patients allocated to the remimazolam group will receive intravenous infusion of remimazolam at a rate of 6 mg/kg/h, followed by 1 mg/kg/h after the loss of consciousness. The infusion rate of remimazolam will be adjusted to a maximum rate of 2 mg/kg/h to achieve a bispectral index of 40 to 60.
  Other Names: Remimazolam Besylate
  Arms: Remimazolam
Drug: Propofol — For the induction of anesthesia, patients allocated to the propofol group will receive a bolus dose of propofol 1.5 mg/kg. After the loss of consciousness, general anesthesia will be maintained with sevoflurane to achieve a bispectral index of 40 to 60.
  Arms: Propofol
Drug: Rocuronium — After the loss of consciousness, a bolus of rocuronium 1 mg/kg was intravenously administered. After 90 seconds of manual ventilation, endotracheal intubation was performed
Drug: Sufentanil — During the study period, a total dose of sufentanil 0.5-2.0 mcg/kg was intravenously administered at the attending anesthesiologists' discretion.

SUMMARY:
Remimazolam is a novel ultra-short-acting benzodiazepine. Several studies demonstrated that its efficacy as a sedative hypnotics for general anesthesia is non-inferior to propofol. However, evidence on the hemodynamic stability of remimazolam for the anesthesia induction in patients undergoing coronary artery bypass grafting is lacking. This prospective randomized trial aims to compare hemodynamic stability during anesthesia induction between remimazolam and propofol in patients undergoing coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (aged 19 years or older) who scheduled for elective coronary artery bypass grafting

Exclusion Criteria:

* Patients who refuse to participate
* Concomitant heart valve surgery or thoracic aorta surgery
* Emergent surgery
* Preoperative sedation
* Intubated state
* Patients with mechanical circulatory assist device
* Preoperative use of inotropes or vasopressors
* History of allergy or adverse reaction to study drugs
* Rapid sequence intubation
* Lactose intolerance
* Peanut allergy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
MAP-time integral | During 10 minute from the administration of the study drug
  The area under the baseline MAP (sec * mmHg). Baseline MAP was defined as the mean MAP over the 3 min period immediately before induction.

SECONDARY OUTCOMES:
Time to loss of consciousness | During 10 minute from the administration of the study drug
  The time from the study drug administration to loss of consciousness
Mean blood pressure | During 10 minute from the administration of the study drug
  maximum / minimum value (mmHg)
Heart rate | During 10 minute from the administration of remimazolam or propofol
  maximum / minimum / mean / median / time-weighted average values (bpm)
Regional cerebral oxygen saturation | During 10 minute from the administration of the study drug
  continuous monitoring of regional cerebral oxygen saturation during surgery (%)
Cardiac output | During 10 minute from the administration of the study drug
  continuous monitoring of cardiac output (L/min)
Sufentanil dose | During 10 minute from the administration of the study drug
  Total dose of administered sufentanil (mcg)
Crystalloid | During 10 minute from the administration of the study drug
  Total volume of administered crystalloid (ml)
Study drug dose | During 10 minute from the administration of the study drug
  Total dose of administered remimazolam or propofol (mg)
Number of vasopressor administration | During 10 minute from the administration of the study drug
  1. Total number (n)
  2. Ephedrine (n)
  3. Phenylephrine (n)
  4. Vasopressin (n)
  5. Norepinephrine (n)
Ephedrine dose | During 10 minute from the administration of the study drug
  Total dose of administered ephedrine (mg)
Phenylephrine dose | During 10 minute from the administration of the study drug
  Total dose of administered phenylephrine (mcg)
Vasopressin dose | During 10 minute from the administration of the study drug
  Total dose of administered vasopressin (unit) 2. Ephedrine: total dose / number of administration 3. Phenylephrine: total dose / number of administration 4. Vasopressin: total dose / number of administration 5. Norepinephrine: total dose / number of administration
Norepinephrine dose | During 10 minute from the administration of the study drug
  Total dose of administered norepinephrine (mcg)

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No